CLINICAL TRIAL: NCT03397875
Title: Effect of Various Sealers on Healing of Teeth With Apical Periodontitis: A Clinical Study
Brief Title: Effect of Various Sealers on Healing of Teeth With Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aparna Tripathi
Record Dates: First submitted 2017-12-31; First posted 2018-01-12 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-04

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — epoxy resin-based root canal sealer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Zinc oxide based sealer (Active Comparator): After root canal treatment obturation with gutta percha will be done using zinc oxide based sealer.
  Interventions: Procedure: Zinc oxide based sealer
- Epoxy resin based sealer (Experimental): After root canal treatment obturation with gutta percha will be done using epoxy resin based sealer.
  Interventions: Procedure: Epoxy resin based sealer
- Bioactive silicone based sealer (Experimental): After root canal treatment obturation with gutta percha will be done using bioactive silicone based sealer.
  Interventions: Procedure: Bioactive silicone based sealer

INTERVENTIONS:
Procedure: Zinc oxide based sealer — After root canal treatment obturation will be done using zinc oxide eugenol based sealer.
  Arms: Zinc oxide based sealer
Procedure: Epoxy resin based sealer — After root canal treatment obturation will be done using epoxy resin based sealer.
  Arms: Epoxy resin based sealer
Procedure: Bioactive silicone based sealer
  Other Names: After root canal treatment obturation will be done using bioactive silicone based sealer.
  Arms: Bioactive silicone based sealer

SUMMARY:
This study will compare the effect of three different sealers on healing of teeth with apical periodontitis after primary root canal treatment.

DETAILED DESCRIPTION:
Various sealers with different chemical composition and properties are available but it is yet not clear if one sealer is superior to other in terms of healing of apical periodontitis.

Three different groups of sealers will be used- a zinc oxide based sealer, an epoxy resin based sealer and a bioactive silicone based sealer. Mature mandibular permanent molar with the diagnosis of apical periodontitis (as confirmed clinically & by periapical radiograph) will be chosen for the study. Primary non surgical root canal treatment will be performed. The sealer will be randomly selected just before obturation of root canals. The patient will be allotted to one of the three groups.

* Group I: Zinc oxide eugenol sealer group. The material will be mixed according to manufacturer instructions and applied to canals using a lentulospiral and the obturation will be performed.
* Group II: Epoxy resin based sealer group. The material will be mixed according to the manufacturer's instructions and obturation will be done.
* Group III: Bioactive silicone based sealer: The material will be used according to the manufacturer's instruction and obturation will be performed

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria of the study will include:

* Patient willing to participate in the study.
* Age >18 years.
* No history of antibiotic use within the past month or requiring antibiotic premedication
* No history of prior analgesic use during past 24 hrs.
* Mature permanent mandibular molar having apical periodontitis requiring primary root canal treatment.
* There must be a radiographic evidence of periapical radiolucency (minimum size 2mmx2mm) and a diagnosis of pulpal necrosis, as confirmed by negative response to cold and electrical tests; and absence of bleeding on entering the pulp chamber

Exclusion Criteria:

* Re-treatment
* Unwillingness of patients
* The presence of a difficult canal anatomy (root canals with an extreme curvature ≥30 deg), internal or external resorption and immature teeth.
* Accident or complication during treatment (calcified canals ,inability to achieve apical patency in any canals) Immuno-compromised, diabetic, pregnant and hypertensive patients.
* Teeth that are peridontally compromised

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Radiographic success | 12 months
  Change in apical bone density will be measured by Periapical Index (PAI) score. PAI score equal to or less than 2 will be categorized as success.
Clinical success | 12 months
  Absence of pain, sinus tract, swelling and mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No